CLINICAL TRIAL: NCT02448082
Title: The Efficacy of Sodium Shale Oil Sulponate 1% Shampoo in the Treatment of Pityriasis Capitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Johannesburg (Other)
Responsible Party: Principal Investigator, Dr J. Pellow, Dr Neil Gower, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ZeenatMia201001496
Record Dates: First submitted 2015-05-04; First posted 2015-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Dandruff
Keywords: Dandruff; Pityriasis capitis; Ichthyol® Pale; Sodium shale oil sulponate 1%
MeSH Terms: conditions — Dandruff

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shampoo (inactive) (Placebo Comparator): Shampoo containing no active anti-dandruff ingredients will be used to wash the participants' hair every second day, starting from day 1 to day 15. Each participant in the placebo group will wash their hair with 25ml of the placebo shampoo per hair washing session.
  Interventions: Other: Shampoo (inactive)
- Sodium shale oil sulponate 1% shampoo (Experimental): Shampoo containing sodium shale oil sulponate 1% will be used to wash the participants' hair every second day, starting from day 1 to day 15. Each participant in the experimental group will wash their hair with 25ml of the sodium shale oil sulponate 1% shampoo per hair washing session.
  Interventions: Other: Sodium shale oil sulponate 1% shampoo

INTERVENTIONS:
Other: Shampoo (inactive) — Shampoo which is made to look and feel the same as the experimental shampoo but does not contain the active ingredient of sodium shale oil sulponate 1%.
  Arms: Shampoo (inactive)
Other: Sodium shale oil sulponate 1% shampoo — Shampoo containing the active ingredient of sodium shale oil sulponate 1%.
  Other Names: Ichthyol® Pale
  Arms: Sodium shale oil sulponate 1% shampoo

SUMMARY:
Dandruff, also known as Pityriasis capitis, is a common condition which affects the scalp of almost half the post-pubertal population regardless of race and gender. It is said that dandruff affects at least 50% of the world's adult population and about 15 - 20% of the world's total population. Dandruff is usually marked by flaking as well as itching and irritation of the scalp which can also lead to greasiness. Dandruff can lead to physiological and psychological issues and can be very distressing and embarrassing for the sufferer, causing low self esteem and social problems. Current treatment options for dandruff include many over-the-counter preparations, anti-dandruff shampoos and topical steroid applications which are accompanied by numerous adverse effects. According to Lunar Pharmaceuticals Ichthyol® Pale is a sodium salt of pale sulphonated shale oil in aqueous solution with anti-microbial properties which can combat dandruff helping with the causative and symptomatic relief of this condition.

The aim of the study is to determine the efficacy of Sodium Shale Oil Sulponate 1% shampoo in the treatment of Pityriasis capitis. This will be evaluated using the Adherent Scalp Flaking Score (ASFS) grading and the Visual Analogue Scale (VAS).

DETAILED DESCRIPTION:
The research study will be performed as a 16 day double-blind placebo controlled study design. The research will be conducted at the University of Johannesburg, Doornfontein Campus. Forty participants, both males and females, between the ages of 18 and 45 years will be recruited via advertisements placed at the University of Johannesburg Health Clinic, Doornfontein Campus, at hair salons and gyms situated around Gauteng (with relevant permission given).

The initial consult (day zero) will consist of a full description and discussion of the research method with the participant. Thereafter, the participant will be requested to read a participant information form and sign a consent form. An evaluation, based on the inclusion and exclusion criteria, to determine whether the participant meets the criteria for the research study will be performed. A physical and general assessment will be conducted to determine vital signs and health status respectively. Thereafter, the participant's dandruff will be evaluated using the Adherent Scalp Flaking Score (ASFS) grading, completed by the researcher, and the Visual Analogue Scale (VAS), completed by both the participant and the researcher.

The participants will be divided into two groups by means of match pairing, according to severity of dandruff. Based on the determined group, the participants will be given either the experimental (with active anti-dandruff agents) or control (without active anti-dandruff agents) shampoo together with the directions for the use of the shampoo at the first consultation. At the second consultation, which will occur on day 8, the participant's scalp will be evaluated using the ASFS grading, completed by the researcher, and the VAS, completed by both the participant and the researcher. On day 16 (final consult), a final evaluation of the participant's dandruff will be done, using the same method described as with the second consultation. At each consult, all results will be recorded. Participants will be requested to wash the scalp once every second day, starting from day 1 to day 16. Reminders to wash the scalp will be sent to each participant via a text message the night before they are due to wash their hair.

On completion of the study, all data will be collated and an Exploratory Data Analysis (EDA) will be performed to determine group normality and comparability of the data. Parametric intergroup analysis will include the independent T-sample test, followed by intragroup analysis using the ANOVA measurement. Non-parametric intergroup analysis will include the Mann-Whitney U test, while intragroup analysis will involve the Friedman or the Wilcoxon Signed-Ranks test.

Positive results of the study may yield an effective and safe treatment option for dandruff.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 45;
* suffering from mild to moderate dandruff with itching, flaking, greasiness, irritation of the scalp and possible hair loss;
* have a baseline Adherent Scalp Flaking Score grading ASFS score of ≥ 24 and 7, and
* have good general health.

Exclusion Criteria:

* Suffering from other conditions such as psoriasis, atopic dermatitis, contact dermatitis or tinea capitis;
* diagnosed with systemic or chronic diseases;
* pregnant or lactating;
* currently on any chronic medication, or
* currently on treatment for dandruff.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Adherent Scalp Flaking Score (ASFS) | 16 days.
  The Adherent Scalp Flaking Score will be conducted by the researcher on days 1,8 and 16.

SECONDARY OUTCOMES:
Dandruff severity as measured by the Visual Analogue Scale (VAS) | 16 days.
  Dandruff severity as measured by the Visual Analogue Scale will be scored by both the researcher and participant on days 1, 8 and 16.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Gower, M.TechHom, Study Director — University of Johannesburg
Locations (1):
- University of Johannesburg, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No